CLINICAL TRIAL: NCT05015387
Title: Efficacy of Proanthocyanidins in Non-Surgical Periodontal Therapy: a Randomized Controlled Trial
Brief Title: Efficacy of Proanthocyanidins in Non-Surgical Periodontal Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Evelina Vedlugaite, Assistant, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Proanthocyanidins
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Periodontitis, Adult
MeSH Terms: conditions — Chronic Periodontitis | interventions — Proanthocyanidins

STUDY DESIGN:
Intervention Model Description: All patients were allocated by the same examiner to two groups: the first group received minimally invasive non-surgical therapy only (MINST group), the second group- minimally invasive non-surgical therapy and subgingival application of collagen hydrogels with PACNs (MINST+PACNs group). The same examiner performed the coding and randomization of the participants in the treatment groups with a computer-generated randomization table.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients were allocated by the Examiner 1. The same examiner performed the coding and randomization of the participants in the treatment groups with a computer-generated randomization table. Both groups received full-mouth minimally invasive non-surgical therapy procedure by single periodontist (Examiner 2), and patients in MINST+PACNs group received collagen hydrogel chips with proanthocyanidins, placed subgingivally in periodontal pockets with PPD≥4mm. After minimally invasive non-surgical therapy patients returned for the next appointment (8 weeks after baseline). Periodontal reevaluation of encoded patients was performed by a single periodontist (Examiner 2).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MINST group (Active Comparator): Patients with periodontitis received minimally invasive non-surgical therapy .
  Interventions: Procedure: Minimally invasive non-surgical therapy; Diagnostic Test: Collection of saliva samples
- MINST+PACNs group (Experimental): Patients with periodontitis received minimally invasive non-surgical therapy and subgingival application of collagen hydrogels with proanthocyanidins.
  Interventions: Procedure: Minimally invasive non-surgical therapy; Combination Product: Subgingival application of collagen hydrogels with proanthocyanidins; Diagnostic Test: Collection of saliva samples

INTERVENTIONS:
Procedure: Minimally invasive non-surgical therapy — Under local anesthesia subgingival instrumentation with ultrasonic and hand instruments and magnification (4.5x) was performed.
Combination Product: Subgingival application of collagen hydrogels with proanthocyanidins — Patients received collagen hydrogel chips with proanthocyanidins from Pelargonium sidoides root extract, placed subgingivally in periodontal pockets with PPD≥4mm after minimally invasive non-surgical therapy.
  Arms: MINST+PACNs group
Diagnostic Test: Collection of saliva samples — For MMP-3/TIMP-1 detection, the collection of saliva samples was performed using Salivette (SARSTEDT AG and Co, Germany) saliva sample collection kit. Saliva samples were collected at the baseline for all patients and 8 weeks after treatment. Samples were centrifuged at 3500 rpm (2 min), aliquoted and protease inhibitors cocktail (1 mg/ml) was added to each sample. All samples were stored at -80oC. MMP-3, TIMP-1 concentration in saliva samples was examined using commercial ELISA kits (Elabscience, USA) and Multiskan Microplate Photometer (Thermo Fisher Scientific) at 450 nm wavelength. Saliva MMP-3/TIMP-1 samples were collected before treatment and 8 weeks after treatment.

SUMMARY:
The aim of the study is to evaluate the efficacy of proanthocyanidins as an adjunctive periodontal therapy in patients with periodontitis. Recently proanthocyanidins were proposed as a viable adjunct to periodontal treatment. Preclinical studies have shown high antibacterial and anti-inflammatory capacities of proanthocyanidins, that could reduce periodontal inflammation and promote periodontal tissues regeneration. In addition, proanthocyanidins demonstrate a specific antibacterial characteristic to attack periodonto-pathogenic bacteria (Porphyromonas gingivalis) but save the oral commensal bacteria (Streptococcus salivarius). Patients with periodontitis (stage III-IV) were included in this study. Patients with periodontitis received two different treatment modalities: minimally invasive non-surgical therapy only (MINST group) or minimally invasive non-surgical therapy and subgingival application of collagen hydrogels with proanthocyanidins (MINST+PACNs group). Clinical periodontal parameters (PPD, CAL, BOP, PI) were evaluated before treatment and after 8 weeks. Concentrations of immunological markers MMP-3 and TIMP-1 in saliva were investigated.

DETAILED DESCRIPTION:
Ethical permission was issued by the Regional Biomedical Research Ethics Committee (No. BE-2-38). All included patients must have signed an informed consent form, were willing and able to show up for follow-up appointments and agreed to coded data collection. Patients were given enough time to analyze protocol of the study and were free to exit the study at any time without a specific reason. The study was performed according to CONSORT guidelines for randomized controlled clinical trials.

Patients with periodontitis (stage III-IV) were included in the study. The inclusion criteria in treatment groups were systemically healthy patients with stage III and IV periodontitis with slow or moderate rate of progression (A/B) (radiographic bone loss extending to middle or apical third of the root, tooth loss due to periodontitis, maximum probing depth≥6mm, horizontal and vertical (≥3mm) bone loss).

All patients were allocated by the Examiner 1 to two groups: the first group received minimally invasive non-surgical therapy only (MINST group), the second group- minimally invasive non-surgical therapy and subgingival application of collagen hydrogels with PACNs (MINST+PACNs group). The same Examiner 1 performed the coding and randomization of the participants in the treatment groups with a computer-generated randomization table.

Clinical trial protocol included several appointments. At the baseline all patients received periodontal examination by periodontist (Examiner 2), the collection of saliva samples was performed. Both groups received full-mouth minimally invasive non-surgical therapy procedure by single periodontist (Examiner 2). During the MINST procedure the periodontist (Examiner 2) was not informed about the patient 's assignment to the group (MINST or MINST+PACNs). After the procedure patient 's allocation to the group was revealed to periodontist by Examiner 1 and accordingly the patient received adjunctive treatment (in MINST+PACNs group received collagen hydrogel chips with proanthocyanidins) or ended the procedure without adjunctive therapy (MINST group). Postoperative care instructions were given (no flossing or use of chemical control materials).

After the procedure patients returned for the next appointment (8 weeks after baseline). Periodontal reevaluation of encoded patients was performed by a single periodontist (Examiner 2). Saliva sample were collected in the same manner as mentioned before.

The relationship of clinical periodontal parameters and MMP-3 and TIMP-1 levels were analyzed to assess the efficacy of proanthocyanidins in periodontal therapy.

The statistical analysis was performed with IBM SPSS 28 (Armonk, NY: IBM Corp.) statistic software package. Shapiro-Wilk test was performed to assess if clinical periodontal measures (per-patient PPD, CAL, BOP and PI) and biochemical measures (MMP-3 and TIMP-1 concentrations in saliva) followed a normal distribution. Accordingly, if the data followed a normal distribution, paired-samples t-test was done to obtain before and after treatment comparisons within the groups. If the assumption of normality was violated, related samples Wilcoxon signed ranks test was done to obtain before and after treatment comparisons within the groups. The between group comparisons of measures were determined by either independent samples t-test in case the specific measure followed a normal distribution or Mann-Whitney test in case the specific measure followed a non-normal distribution. The statistical significance level was considered at the 0.05 level.

ELIGIBILITY:
Inclusion criteria:

* patients with stage III and IV periodontitis with slow or moderate rate of progression (A/B) (radiographic bone loss extending to middle or apical third of the root, tooth loss due to periodontitis, maximum probing depth≥6mm, horizontal and vertical (≥3mm) bone loss);
* systemically healthy individuals;
* have≥ 20 remaining teeth;
* ≥30 years patients.

Exclusion criteria:

* patients with stage I and II periodontitis (radiographic bone loss in coronal third, no tooth loss due to periodontitis, maximum probing depth ≤5mm, mostly horizontal bone loss);
* patients with systemic diseases;
* had antibiotic therapy during the last 3 months;
* had periodontal treatment during last 6 months;
* were pregnant or lactating women;
* claimed to be allergic to the adjunct (proanthocyanidins).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Mean PPD change from baseline in moderate sites at 8 weeks | Before treatment and 8 weeks after baseline
  Pocket probing depth is measured with periodontal probe. Pocket probing depth from gingival margin to the bottom of periodontal pocket.

SECONDARY OUTCOMES:
Mean PPD change from baseline in deep sites at 8 week | Before treatment and 8 weeks after baseline
  Pocket probing depth is measured with periodontal probe. Pocket probing depth from gingival margin to the bottom of periodontal pocket.
Mean CAL changes from baseline at 8 week | Before treatment and 8 weeks after baseline
  Clinical attachment level is measured with periodontal probe.
Mean PI changes from baseline at 8 week | Before treatment and 8 weeks after baseline
  Presence or absence of plaque is measured.
Mean BOP change from baseline in deep sites at 8 week | Before treatment and 8 weeks after baseline
  Presence or absence of bleeding during periodontal probing.
Mean MMP-3, TIMP-1 changes from baseline at 8 week | Before treatment and 8 weeks after baseline
  Biomarkers MMP-3 (matrix metalloproteinase-3) and TIMP-1 (endogenous tissue inhibitors of metalloproteinases-1) concentration in salivary samples.

CONTACTS AND LOCATIONS:
Overall Officials: Nijolė Savickienė, PhD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Jekabsone A, Sile I, Cochis A, Makrecka-Kuka M, Laucaityte G, Makarova E, Rimondini L, Bernotiene R, Raudone L, Vedlugaite E, Baniene R, Smalinskiene A, Savickiene N, Dambrova M. Investigation of Antibacterial and Antiinflammatory Activities of Proanthocyanidins from Pelargonium sidoides DC Root Extract. Nutrients. 2019 Nov 19;11(11):2829. doi: 10.3390/nu11112829. PMID 31752295
- [Background] Savickiene N, Jekabsone A, Raudone L, Abdelgeliel AS, Cochis A, Rimondini L, Makarova E, Grinberga S, Pugovics O, Dambrova M, Pacauskiene IM, Baseviciene N, Viskelis P. Efficacy of Proanthocyanidins from Pelargonium sidoides Root Extract in Reducing P. gingivalis Viability While Preserving Oral Commensal S. salivarius. Materials (Basel). 2018 Aug 22;11(9):1499. doi: 10.3390/ma11091499. PMID 30135370